CLINICAL TRIAL: NCT02345577
Title: Effects of Stochastic Whole-body Vibration Physiotherapy-WBV (Stochastic Resonance Physiotherapy-SRT) on Muscle Strength in Patients After Kidney Transplantation: a Pilot Study
Brief Title: Whole-body Vibration Physiotherapy in Kidney Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruitment rate
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 176/14
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Stochastic whole body vibration therapy; Muscle strength; Intramuscular lipid content; Intramyocellular lipid content; Short Physical Performance Battery Test; Prospective, randomised , double blind,placebo-controlled trial; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapeutical intervention (Active Comparator): 3 WBV-sessions per week for 3 consecutive months. Each session consists of 5 series with a duration of 60 sec with 60 sec rest-time with vibration of increasing frequency starting at 1Hz / Noise 4 going up to 6Hz / Noise 5 depending on patients' tolerability and with a fixed 3mm amplitude.
  Interventions: Other: Stochastic whole body vibration (WBV) therapy - Physiotherapeutical intervention
- Sham physiotherapeutical intervention (Sham Comparator): 3 WBV-sessions per week for 3 consecutive months. Each session consists of 5 series with a duration of 60 sec with 60 sec rest-time at 1 Hz / Noise 1 and 3mm amplitude.
  Interventions: Other: Stochastic whole body vibration (WBV) therapy - Sham physiotherapeutical intervention

INTERVENTIONS:
Other: Stochastic whole body vibration (WBV) therapy - Physiotherapeutical intervention — Physiotherapeutical intervention
  Arms: Physiotherapeutical intervention
Other: Stochastic whole body vibration (WBV) therapy - Sham physiotherapeutical intervention — Sham physiotherapeutical intervention
  Arms: Sham physiotherapeutical intervention

SUMMARY:
Kidney recipients loose significant amounts of muscle mass and skeleton minerals in the early post-transplantation period and suffer from increasing abnormalities of neuromuscular functions.

Stochastic whole body vibration (WBV) therapy is a relatively new form of movement physiotherapy that is used for strength training. Various clinical studies have shown that in addition to muscle function, WBV also improved body balance and bone mineral density. To study the impact of stochastic WBV physiotherapy on musculoskeletal parameters after renal transplantation, kidney transplant recipients will be enrolled and undergo WBV. The investigators hypothesize that WBV physiotherapy improves both maximum muscle strength and muscular performance

DETAILED DESCRIPTION:
Background

The increasing incidence of muscular wasting, bone disease, falls and related fractures are the price for excellent survival rates in transplanted patients. Kidney recipients loose significant amounts of muscle mass and skeleton minerals in the early post-transplantation period and suffer from increasing abnormalities of neuromuscular functions.

Recently, stochastic whole-body vibration (WBV) has received much attention as a potential muscle-anabolic and anti-osteoporotic intervention. It is suggested that the randomized low-frequency signals produced during such training can activate otherwise high threshold afferent and efferent motor-neurons and thus may result in a considerable neuromuscular activation. Additionally, there data supporting peripherally-induced central biochemical activation, that meaning the production of CNS modulators due to application of mechanical exercise such as stochastic WBV. The result is a rapid (within minutes), transient force increase. Due to the high number of stimuli-repetitions, it is possible to increase muscle strength using shorter training times (<5 min) than with conventional physiotherapeutic methods (> 30 min). Several experimental and clinical studies have shown that in addition to muscle function, WBV also improved body balance and bone mineral density.

Moreover, a population of renal transplant recipients has not yet been studied elsewhere.

WBV is a very appealing approach, foremost in subjects with limited physical activity; it represents a potentially simple and efficient training method for skeletal muscle and better functional performance, thus preventing falls and consequently fractures.

Objective

Primary:

- To determine the effect of post-transplantation stochastic WBV therapy on preservation of functional muscle strength.

Secondary:

To assess a) the efficacy of post-transplantation stochastic WBV on body balance b) the efficacy of post-transplantation stochastic WBV on preservation of lean muscle mass determined by Magnetic Resonance Spectroscopy (MRS) c) the changes in bone turnover markers in renal transplant recipients under stochastic WBV therapy d) the short-term safety of stochastic WBV therapy in renal transplant recipients.

Methods

Prospective, randomized, double-blinded, placebo-controlled setting.

Recruited individuals will be randomized in Group 1 (intervention) and in Group 2 (placebo). All participants will be evaluated monthly for occurrence of falls and fractures, and treatment-associated side effects. Testing will be performed upon study entry and at 3 and 6 months according to the following schedule:

Visit 1 (Baseline):

* Muscle strength measurement
* Neuromuscular tests (SPPBT)
* Magnetic resonance spectroscopy (MRS)
* Turnover Markers (blood) Visits 2 and 3 (after 3 and 6 months respectively): Identical to visit 1

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Kidney transplantation in the last 12 months
* Stable kidney function (eGFR>20 ml/min)
* No episode of acute rejection during the last 2 months
* Written informed consent

Exclusion Criteria

* Inability to posture or to perform whole-body vibration therapy or MRS after transplantation
* Treatment with anabolic medication, fluorine, bisphosphonates, or hormone replacement therapy (estrogens, selective modulators of the estrogenic receptors) within the previous 3 months
* Treatment with high-dose steroid therapy due to acute rejection episode during the last 2 months before study inclusion
* Implanted devices (pacemakers, defibrillators, stents, etc.)
* Pregnancy
* Previous ophthalmic cataract surgery
* Previous history of epilepsy
* Previous recent spine of leg fracture (last 3 months)
* Other individuals especially in need of protection (according to the Swiss Academy of Medical Sciences)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Change in maximal isometric strength of the leg extensors from baseline to 3 and 6 months | 6 months

SECONDARY OUTCOMES:
Change of neuromuscular test (SPPBT)-score from baseline to 3 and 6 months | 6 months
Change of muscle mass from baseline to 3 and 6 months | 6 months
Change of intramuscular lipid content from baseline to 3 and 6 months | 6 months
Change of intramyocellular (calf) lipid content from baseline to 3 and 6 months | 6 months
Falls during study period | 6 months
Fractures during study period | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Spyridon Arampatzis, MD, Principal Investigator — Department of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital
Locations (1):
- Department of Nephrology, Hypertension and Clinical Pharmacology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Streja E, Molnar MZ, Kovesdy CP, Bunnapradist S, Jing J, Nissenson AR, Mucsi I, Danovitch GM, Kalantar-Zadeh K. Associations of pretransplant weight and muscle mass with mortality in renal transplant recipients. Clin J Am Soc Nephrol. 2011 Jun;6(6):1463-73. doi: 10.2215/CJN.09131010. Epub 2011 Mar 17. PMID 21415312
- [Background] Lai CL, Tseng SY, Chen CN, Liao WC, Wang CH, Lee MC, Hsu PS. Effect of 6 months of whole body vibration on lumbar spine bone density in postmenopausal women: a randomized controlled trial. Clin Interv Aging. 2013;8:1603-9. doi: 10.2147/CIA.S53591. Epub 2013 Dec 4. PMID 24348029
- [Background] Rogan S, Hilfiker R, Schmid S, Radlinger L. Stochastic resonance whole-body vibration training for chair rising performance on untrained elderly: a pilot study. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):468-73. doi: 10.1016/j.archger.2012.02.011. Epub 2012 Mar 16. PMID 22425243
- [Background] Rogan S, Hilfiker R, Herren K, Radlinger L, de Bruin ED. Effects of whole-body vibration on postural control in elderly: a systematic review and meta-analysis. BMC Geriatr. 2011 Nov 3;11:72. doi: 10.1186/1471-2318-11-72. PMID 22054046
- [Background] Calendo LR, Taeymans J, Rogan S. [Does muscle activation during whole-body vibration induce bone density improvement in postmenopausal women?--A systematic review]. Sportverletz Sportschaden. 2014 Sep;28(3):125-31. doi: 10.1055/s-0034-1366545. Epub 2014 May 14. German. PMID 24828509